CLINICAL TRIAL: NCT01680952
Title: Study to Evaluate the Safety and Efficacy of Extended Release Tacrolimus (Advagraf®) + Sirolimus (Rapamune®), Versus Extended Release Tacrolimus (Advagraf®) + Mycophenolate Mofetil in Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0920
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Transplant Patients
Keywords: RECORD study
MeSH Terms: interventions — Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A) TEST (Active Comparator)
  Interventions: Drug: A) TEST; Drug: B) CONTROL
- B) CONTROL (Experimental)
  Interventions: Drug: A) TEST; Drug: B) CONTROL

INTERVENTIONS:
Drug: A) TEST — 1. Extended Release Tacrolimus (Advagraf®)
     ① Living The day before surgery: 0.2 mg/kg(morning dose) po, qd Morning on the day of surgery: 0.1 mg/kg po, qd After surgery, the capacity is adjusted according to the trough level. clinical significance, electrolyte level.
     ② Cadaveric Before surgery at once : 0.1 mg/kg within 12hours before surgery. After surgery : 0.2mg/kg po. in the morning After that, the capacity is adjusted according to the trough level. clinical significance, electrolyte level.
  2. Sirolimus (Rapamune®):
  After surgery : 2mg/kg po. within 24hrs after reperfusion. After that, the capacity is adjusted according to the trough level.
  Other Names: 1. Test group : Extended Release Tacrolimus (Advagraf®) + Sirolimus (Rapamune®)
Drug: B) CONTROL — 1. Extended Release Tacrolimus (Advagraf®)
     : Same as above.
  2. Mycophenolate mofetil : After surgery : 500mg/kg po. within 24hrs after reperfusion. After that, daily dose: 1000mg bid
  Other Names: 2. Control group: Extended Release Tacrolimus (Advagraf®) + Mycophenolate mofetil

SUMMARY:
This study will compare the efficacy and safety of Extended Release Tacrolimus (Advagraf®) + Sirolimus (Rapamune®), versus Extended Release Tacrolimus (Advagraf®) + Mycophenolate mofetil in Kidney Transplant Patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged over 20 years
* Patient who is judged would have the benefits of the Extended Release Tacrolimus (Advagraf®)treatment by the investigator
* Patients has given written informed consent
* Patient is a recipient of primary or recipient of primary (a living kidney transplant, a cadaveric donor.)
* Patients has received an ABO compatible donor kidney.
* Complement-dependent Cytotoxic Crossmatch: CDC) result: negative
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within 7 days prior to enrollment or upon hospitalization

Exclusion Criteria:

* Patient has previously received an organ transplant other than a kidney.
* Patient has a known hypersensitivity to tacrolimus, Sirolimus (Rapamune®),Mycophenolate mofetil.
* Desensitization
* HLA-identical
* Heart Disease; Heart failure (symptom, EF <45%)
* Lung Disease; Significant chronic obstructive pulmonary disease, restrictive lung disease
* Patient has an uncontrolled concomitant infection (including Hepatitis B, Hepatitis C) or any other unstable
* malignant tumor history in the 5years prior to enrollment. (except,squamous cell carcinoma)
* Patient has received a kidney transplant from non-heart beating donor
* Cold ischemic time > 30hrs
* Elevated AST and/or ALT levels greater than 3 times the upper value of the normal range of the investigational site
* (ANC)<1,500/mm3, (WBC)<2,500/ mm3, (PLT)<100,000/ mm3
* ATG: Anti-thymocyte globulin induction
* Medical condition that could interfere with the study objectives.
* Patient is currently taking or has been taking an investigational products in the 30 days prior to enrollment.
* Patient is currently taking or has been taking an prohibited medications in the 28 days prior to enrollment.
* Patient who is judged not to be adequate by the investigator owing to other reasons
* Patient is pregnant or lactating.
* Recipient or donor is known to be seropositive for human immunodeficiency virus.(HIV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Failure rate in effectiveness of up to 12 months after kidney transplant | 12 months after kidney transplant
  1. Biopsy confirmed acute rejection
  2. Subjects and graft survival
  3. Glomerular filtration rate (GFR)
  4. 24-hour urine test results at 12 months after kidney transplant: Urine protein, CrCl.

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Kyungpook national hospital, Daegu, Daegu
  - Ajou Univeristy Medical Center, Suwon, KyungKi Province
  - Severance hospital, Seoul, Seoul
  - Gangnam Severance hospital, Seoul, Seoul
  - Korea University Anam Hospital, Seoul, Seoul
  - Seoul National University hospital, Seoul, Seoul
  - Ulsan Univ Hospital, Ulsan, Ulsan

REFERENCES:
- [Derived] Huh KH, Lee JG, Ha J, Oh CK, Ju MK, Kim CD, Cho HR, Jung CW, Lim BJ, Kim YS; RECORD Study. De novo low-dose sirolimus versus mycophenolate mofetil in combination with extended-release tacrolimus in kidney transplant recipients: a multicentre, open-label, randomized, controlled, non-inferiority trial. Nephrol Dial Transplant. 2017 Aug 1;32(8):1415-1424. doi: 10.1093/ndt/gfx093. PMID 28810721